CLINICAL TRIAL: NCT01696604
Title: A Single-center, Randomized, Blinded, Placebo-controlled Two-part Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of the Selective Androgen Receptor Modulator (SARM), GSK2849466, in Single and Repeat Doses, With and Without Food, in Healthy Male Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GSK2849466 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 116715
Record Dates: First submitted 2012-09-27; First posted 2012-10-01 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Cachexia
Keywords: safety; pharmacokinetics; FTIH; SARM
MeSH Terms: conditions — Cachexia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- Part A: Cohort 1-GSK2849466 (Experimental): The subjects will receive single planned dose of GSK284946 in ascending order (0.01, 0.03, 0.1, and 0.3 mg) in ratio of 3:1.with placebo within each of 4 treatment periods. The dose will not be allowed to exceed 30 mg over a 24-hour period.
  Interventions: Drug: GSK2849466
- Part A: Cohort 1-Placebo (Experimental): The subjects will receive single dose of matching placebo in one of the 4 treatment periods.
  Interventions: Drug: Placebo
- Part A: Cohort 2-GSK2849466 (Experimental): The subjects will receive single planned dose of GSK284946 in ascending order (0.3, 1, 3, and 10 mg) in ratio of 3:1.with placebo within each of 4 treatment periods. The dose will not be allowed to exceed 30 mg over a 24-hour period in one of the 4 treatment periods.
  Interventions: Drug: GSK2849466
- Part A: Cohort 2-Placebo (Experimental): The subjects will receive single dose of matching placebo in one of the 4 treatment periods.
  Interventions: Drug: Placebo
- Part B: Cohort 3-GSK2849466 (Repeat dose 1) (Experimental): The selection of appropriate doses for Part B will be performed upon consideration of available safety and tolerability and PK data from Part A and/or any preceding repeat dose cohorts. The subjects will receive GSK2849466 in ratio of 3:1.with placebo.
  Interventions: Drug: GSK2849466
- Part B: Cohort 3-Placebo (Repeat dose 1) (Experimental): The subjects will receive repeat dose of matching placebo.
  Interventions: Drug: Placebo
- Part B: Cohort 4-GSK2849466 (Repeat dose 2) (Experimental): The selection of appropriate doses for Part B will be performed upon consideration of available safety and tolerability and PK data from Part A and/or any preceding repeat dose cohorts. The subjects will receive GSK2849466 in ratio of 3:1.with placebo. In Cohort 4 subjects will be dosed in the fasted state on Days 1 and 14 and in the fed state on Day 7.
  Interventions: Drug: GSK2849466
- Part B: Cohort 4-Placebo (Repeat dose 2) (Experimental): The subjects will receive repeat doses of matching placebo.
  Interventions: Drug: Placebo
- Part B: Cohort 5-GSK2849466 (Repeat dose 3) (Experimental): The selection of appropriate doses for Part B will be performed upon consideration of available safety and tolerability and PK data from Part A and/or any preceding repeat dose cohorts. The subjects will receive GSK2849466 in ratio of 3:1.with placebo
  Interventions: Drug: GSK2849466
- Part B: Cohort 5-Placebo (Repeat dose 3) (Experimental): The subjects will receive repeat doses of matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK2849466 — GSK2849466 will be available as capsules of dose strengths 0.01, 0.1, 1.0, and 2.5 mg.
  Arms: Part A: Cohort 1-GSK2849466; Part A: Cohort 2-GSK2849466; Part B: Cohort 3-GSK2849466 (Repeat dose 1); Part B: Cohort 4-GSK2849466 (Repeat dose 2); Part B: Cohort 5-GSK2849466 (Repeat dose 3)
Drug: Placebo — Matching placebo capsules will be available.
  Arms: Part A: Cohort 1-Placebo; Part A: Cohort 2-Placebo; Part B: Cohort 3-Placebo (Repeat dose 1); Part B: Cohort 4-Placebo (Repeat dose 2); Part B: Cohort 5-Placebo (Repeat dose 3)

SUMMARY:
This study is the first administration of GSK2849466 in humans. This will be a single centre, randomized, double-blind, placebo-controlled study, to investigate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of GSK2849466, given as single and repeat oral doses up to 14 days to healthy male subjects. Part A will be a randomized placebo controlled and 4-way crossover study. It will include two cohorts of 8 subjects each. In each cohort there will be 4 study periods each approximately of 1 week including 6 days of washout. Each subject will receive a total of 3 active doses as ascending single oral dose of GSK2849466 and 1 placebo dose during the course of their participation in the study. The first ("bridging dose") dose provided to subjects in Cohort 2 will be the same as the last dose provided to subjects in Cohort 1. The single doses of GSK2849466 planned in Part A of this study are: 0.01, 0.03, 0.1, and 0.3 milligram (mg) in Cohort 1 and 0.3, 1, 3, and 10 mg in Cohort 2. In cohorts 1 and 2 all available safety, tolerability, and PK data will be reviewed prior to each dose escalation. The dosing schedule in Part A may be adjusted to expand a cohort or to add an additional cohort(s) in order to further evaluate additional doses or repeat evaluation of a dose level already studied. Part B will be a randomized placebo controlled, parallel group study. It will include three cohorts of 12 subjects each. Each subject will receive repeat doses of GSK2849466 over 14 days. The doses chosen for Part B will be based on the safety, tolerability, and PK data from Part A. Subjects in Cohort 4 (and/or an another cohort [s] as determined based on Part A PK data) will be dosed in the fasted state on Days 1 and 14 and in the fed state on Day 7 when subjects will receive a standard meal 30 minutes prior to dosing. Part B will provide sufficient safety and tolerability data to bridge to longer duration studies. The study duration, including screening and follow-up, is not expected to exceed 70 days for subjects in the study.

ELIGIBILITY:
Inclusion Criteria:

* Males between 18 and 50 years of age (inclusive), at the time of signing the informed consent form.
* Body weight >=50 kilogram (kg) and Body Mass Index (BMI) within the range 19 - 32 kg/meter (m)^2 (inclusive), where BMI = (weight in kg)/(height in meters)^2.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GlaxoSmithKline (GSK) Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in the Lifestyle Section of the protocol. This criterion must be followed through the completion of the follow-up visit.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Average corrected QT interval using Fridericia's formulas (QTcF) <450 milliseconds (msec); or QTcF <480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

* Subjects with a history of clinically significant endocrine, gastrointestinal, hepatic, cardiovascular, neurological, hematological, immunological, renal, respiratory, or genitourinary abnormalities or diseases.
* Subjects with a history at any time in the past of coronary artery disease, congestive heart failure, angina, myocardial infarction, any cardiac surgery, valvular heart disease, clinically significant arrhythmia, dyspnea, pulmonary edema, stroke, or transient ischemic attack.
* ECG exclusion criteria: Heart rate <40 and >100 beats per minute; PR Interval <120 and >200 msec; QRS duration <70 and >110 msec.
* Subjects with a history of malignancy that is not in complete remission for at least 5 years or 1 year for non-melanoma skin carcinoma.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of drug or alcohol abuse within 5 years prior to the Screening Period.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 grams (g) of alcohol: 12 ounces (360 millilitre [mL]) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor.
* Subjects with a family history of early onset prostate cancer or multiple members with prostate cancer.
* A positive pre-study drug or alcohol screen.
* Cotinine levels indicative of smoking or history or regular use of tobacco-or nicotine-containing products within 6 months prior to screening.
* Subjects with values outside the specified ranges for the following Key Clinical Laboratory Tests must be excluded from the study: Liver function tests - Alanine transaminase (ALT), Direct Bilirubin, or Albumin >10% outside the normal reference range (<0.9 x lower limit of normal [LLN] or >1.1 x Upper Limit of Normal [ULN]), Renal function - Creatinine <1.6 mg/ deciliter (dl) with an age appropriate Glomerular filtration rate (GFR) >=60 mL/min/1.73 m^2), Electrolytes - Sodium > +,- 5 milliequivalents of solute per litre of solvent (mEq/L) outside the normal reference range, Potassium or Calcium >10% outside the normal reference range (<0.9 x LLN or >1.1 x ULN), Metabolic - Glucose >10% outside the normal reference range (<0.9 x LLN or >1.1 x ULN) and Total Cholesterol >240 mg/dl, Muscle - creatine phosphokinase >2.0 x ULN, Hematology - Hemoglobin, WBC, Neutrophils, or Platelets >10% outside the normal reference range (<0.9 x LLN or >1.1 x ULN), Prostate Specific Antigen (PSA) >=2.5 nanogram (ng)/mL.
* A positive test for human immunodeficiency virus (HIV) antibody.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unable to refrain from prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication and throughout the study, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 3 months (12 weeks), 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56-day period.
* Unable to refrain from consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* Unwillingness or inability to follow the procedures outlined in the protocol

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2012-09-26 (Actual); Primary Completion 2013-05-03 (Actual); Study Completion 2013-05-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single ascending doses GSK2849466 as assessed by number of subjects with adverse events (AE)s | 28 days
  Safety and tolerability parameters will include recording of AEs, throughout the study.
Safety and tolerability of repeat doses of GSK2849466 as assessed by number of subjects with AEs | 14 days
  Safety and tolerability parameters will include recording of AEs, throughout the study.
Safety and tolerability of single ascending doses of GSK2849466 as assessed by change from Baseline in electrocardiogram (ECG) readings | 28 days
  Safety and tolerability parameter will include the ECG readings at Baseline and at end of the study.
Safety and tolerability of repeat doses of GSK2849466 as assessed by change from Baseline in ECG readings | 14 days
  Safety and tolerability parameter will include the ECG readings at Baseline and at end of the study.
Safety and tolerability of single ascending doses of GSK2849466 as assessed by change from Baseline in clinical monitoring of blood pressure | 28 days
  Safety and tolerability parameters will include blood pressure readings at Baseline and at end of the study.
Safety and tolerability of repeat doses of GSK2849466 as assessed by change from Baseline in clinical monitoring of blood pressure | 14 days
  Safety and tolerability parameters will include blood pressure readings at Baseline and at end of the study.
Safety and tolerability of single ascending doses of GSK2849466 as assessed by change from Baseline in heart rate | 28 days
  Safety and tolerability parameters will include heart rate at Baseline and at end of the study.
Safety and tolerability of repeat doses of GSK2849466 as assessed by change from Baseline in heart rate | 14 days
  Safety and tolerability parameters will include heart rate at Baseline and at end of the study.
Safety and tolerability of GSK2849466 as assessed by change from Baseline in cardiac telemetry | Part A-Day 1 continuous at least 12 hours post-dose of each dosing session; Part B-Day 1, 4, 7, 10 and 14 continuous at least 8 hours post-dose
  Safety and tolerability parameters will include cardiac telemetry recording at Baseline and at end of the study.
Safety and tolerability of single ascending doses of GSK2849466 as assessed by change from Baseline in laboratory assessments | 28 days
  Safety and tolerability parameters will include laboratory values at Baseline and at end of the study.
Safety and tolerability of repeat doses of GSK2849466 as assessed by change from Baseline in laboratory assessments | 14 days
  Safety and tolerability parameters will include laboratory values at Baseline and at end of the study.

SECONDARY OUTCOMES:
Area under the time-concentration curve from time zero (pre-dose) to last time of quantifiable concentration (AUC(0-t)) and AUC from zero to infinity (AUC(0-inf)) following single doses of GSK2849466 | 2 days of each treatment period in Part A: Day 1-0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 12 hours post dose; Day 2-24 hours post Day 1 dose.
  The AUC(0-t) and AUC(0-inf) for GSK2849466 will be assessed following single doses of GSK2849466.
Maximum concentration (Cmax) following single doses of GSK2849466 | 2 days of each treatment period in Part A: Day 1-0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 12 hours post dose; Day 2-24 hours post Day 1 dose.
  The Cmax of GSK2849466 will be assessed following single doses of GSK2849466.
Time to maximum observed plasma drug concentration (Tmax) following single doses of GSK2849466 | 2 days of each treatment period in Part A: Day 1-0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 12 hours post dose; Day 2-24 hours post Day 1 dose.
  The Tmax for GSK2849466 will be assessed following single doses of GSK2849466.
Terminal half-life (t1/2) following single doses of GSK2849466 | 2 days of each treatment period in Part A: Day 1-0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 12 hours post dose; Day 2-24 hours post Day 1 dose.
  The t1/2 for GSK2849466 will be assessed following single doses of GSK2849466.
The AUC(0-t), AUC(0-inf)) and AUC from time zero to the end of the dosing interval at steady state AUC(0-tau) following repeat doses of GSK2849466 | Part B (all cohorts): Day 1, 2, 14, 15(24 hours serial sampling); Day 4, 5, 6, 7 (pre dose sampling). Part B (Cohort 4): Day 7 and 8 (24 hours serial sampling) and no PK samples on Day 8 if fasted on Day 7.
  The AUC(0-t), AUC(0-inf) and AUC(0-tau) following repeat doses of GSK2849466 with and without food (Cohort 4 and/or another cohort(s) as determined based on Part A PK data) will be assessed in Part B of the study.
The Cmax following repeat doses of GSK2849466 | Part B (all cohorts): Day 1, 2, 14, 15(24 hours serial sampling); Day 4, 5, 6, 7 (pre dose sampling). Part B (Cohort 4): Day 7 and 8 (24 hours serial sampling) and no PK samples on Day 8 if fasted on Day 7.
  The Cmax following repeat doses of GSK2849466 with and without food (Cohort 4 and/or another cohort(s) as determined based on Part A PK data) will be assessed in Part B of the study.
The Tmax following repeat doses of GSK2849466 | Part B (all cohorts): Day 1, 2, 14, 15(24 hours serial sampling); Day 4, 5, 6, 7 (pre dose sampling). Part B (Cohort 4): Day 7 and 8 (24 hours serial sampling) and no PK samples on Day 8 if fasted on Day 7.
  The Tmax following repeat doses of GSK2849466 with and without food (Cohort 4 and/or another cohort(s) as determined based on Part A PK data) will be assessed in Part B of the study.
The t1/2 following repeat doses of GSK2849466 | Part B (all cohorts): Day 1, 2, 14, 15(24 hours serial sampling); Day 4, 5, 6, 7 (pre dose sampling). Part B (Cohort 4): Day 7 and 8 (24 hours serial sampling) and no PK samples on Day 8 if fasted on Day 7.
  The t1/2 following repeat doses of GSK2849466 with and without food (Cohort 4 and/or another cohort(s) as determined based on Part A PK data) will be assessed in Part B of the study.
The estimation of an accumulation ratio following repeat doses of GSK2849466 | Part B (all cohorts): Day 1, 2, 14, 15(24 hours serial sampling); Day 4, 5, 6, 7 (pre dose sampling). Part B (Cohort 4): Day 7 and 8 (24 hours serial sampling) and no PK samples on Day 8 if fasted on Day 7.
  The estimation of an accumulation ratio following repeat doses of GSK2849466 with and without food (Cohort 4 and/or another cohort(s) as determined based on Part A PK data) will be assessed in Part B of the study.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 116715 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116715?search=study&study_ids=116715#rs
- Available data/document: Annotated Case Report Form: 116715 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116715 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116715 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116715 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116715 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116715 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116715 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register